CLINICAL TRIAL: NCT05089084
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of ARO-APOC3 in Adults With Familial Chylomicronemia Syndrome
Brief Title: Study of ARO-APOC3 (Plozasiran) in Adults With Familial Chylomicronemia Syndrome (FCS)
Acronym: PALISADE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-3001
Expanded Access: NCT06796426 (Available)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Familial Chylomicronemia
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — plozasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ARO-APOC3 (Plozasiran) 25 mg (Experimental): Randomized Period: plozasiran 25 mg Q3M for a total of 4 doses.
  Open-label Period (Parts A and B): plozasiran 25 mg Q3M for a total of 8 doses.
  Interventions: Drug: Plozasiran
- Placebo for ARO-APOC3 (Plozasiran) 25 mg (Placebo Comparator): Randomized Period: volume-matched placebo every 3 months (Q3M) for a total of 4 doses.
  Open-label Period (Parts A and B): plozasiran 25 mg Q3M for a total of 8 doses.
  Interventions: Drug: Plozasiran; Drug: Placebo
- ARO-APOC3 (Plozasiran) 50 mg (Experimental): Randomized Period: plozasiran 25 mg Q3M for a total of 4 doses.
  Open-label Period: plozasiran 50 mg (Part A), then 25 mg (Part B) Q3M for a total of 8 doses.
  Interventions: Drug: Plozasiran
- Placebo for ARO-APOC3 (Plozasiran) 50 mg (Placebo Comparator): Randomized Period: volume-matched placebo every 3 months (Q3M) for a total of 4 doses.
  Open-label Period: plozasiran 50 mg (Part A), then 25 mg (Part B) Q3M for a total of 8 doses.
  Interventions: Drug: Plozasiran; Drug: Placebo

INTERVENTIONS:
Drug: Plozasiran — ARO-APOC3 subcutaneous (SC) injection
  Other Names: ARO-APOC3
Drug: Placebo — sterile normal saline (0.9% NaCl) SC injection
  Arms: Placebo for ARO-APOC3 (Plozasiran) 25 mg; Placebo for ARO-APOC3 (Plozasiran) 50 mg

SUMMARY:
The purpose of AROAPOC3-3001 is to evaluate the efficacy and safety of ARO-APOC3 (plozasiran) in adult participants with familial chylomicronemia syndrome (FCS). Participants who have met all eligibility criteria will be randomized to receive 4 doses of plozasiran or matching placebo administered subcutaneously. Participants who complete the randomized period will continue in a 2-year open-label extension period where all participants will receive plozasiran.

ELIGIBILITY:
Inclusion Criteria:

* Fasting triglycerides (TG) ≥ 10 mmol/L (≥ 880 mg/dL) at screening refractory to standard lipid lowering therapy
* Diagnosis of FCS
* Willing to follow dietary counseling as per investigator judgement based on local standard of care
* Participants of childbearing potential (males & females) must use highly-effective contraception during the study and for at least 24 weeks following the last dose of study medication. Males must not donate sperm during the study and for at least 24 weeks following the last dose of study medication
* Women of childbearing potential must have a negative pregnancy test at Screening and cannot be breastfeeding
* Women of childbearing potential on hormonal contraceptives must be stable on the medication for ≥ 2 menstrual cycles prior to Day 1

Exclusion Criteria:

* Current use or use within the last 365 Days from Day 1 of any hepatocyte-targeted siRNA or antisense oligonucleotide molecule
* Diabetes mellitus newly diagnosed within 12 weeks of Screening or where HbA1c ≥ 9.0% at Screening
* Active pancreatitis within 12 weeks before Day 1
* History of acute coronary syndrome event within 24 weeks of Day 1
* History of major surgery within 12 weeks of Day 1
* Uncontrolled hypertension
* On treatment with human immunodeficiency virus (HIV) antiretroviral therapy
* Seropositive for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* New York Heart Association (NYHA) Clas II, III, or IV heart failure

Note: Additional Inclusion/Exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (9):
  - Clinical Site 1, Boca Raton, Florida
  - Clinical Site 2, Suwanee, Georgia
  - Clinical Site 3, Indianapolis, Indiana
  - Clinical Site 4, Elkridge, Maryland
  - Clinical Site 5, St Louis, Missouri
  - Clinical Site 7, New York, New York
  - Clinical Site 6, New York, New York
  - Clinical Site 8, Austin, Texas
  - Clinical Site 9, Norfolk, Virginia
- Argentina (2):
  - Clinical Site 10, Córdoba
  - Clinical Site 11, Formosa
- Australia (5):
  - Clinical Site 14, Camperdown, New South Wales
  - Clinical Site 15, St Leonards, New South Wales
  - Clinical Site 16, Melbourne, Victoria
  - Clinical Site 12, Melbourne
  - Clinical Site 13, Nedlands
- Clinical Site 17, Graz, Austria
- Belgium (4):
  - Clinical Site 18, Edegem
  - Clinical Site 19, Ghent
  - Clinical Site 20, Leuven
  - Clinical Site 21, Liège
- Canada (5):
  - Clinical Site 22, London, Ontario
  - Clinical Site 23, Toronto, Ontario
  - Clinical Site 24, Chicoutimi, Quebec
  - Clinical Site 25, Montreal, Quebec
  - Clinical Site 26, Québec, Quebec
- Clinical Site 27, Zagreb, Croatia
- France (2):
  - Clinical Site 29, Marseille, Cedez 05
  - Clinical Site 28, Paris
- Germany (2):
  - Clinical Site 30, Jena
  - Clinical Site 31, Leipzig
- Clinical Site 32, Galway, Ireland
- Clinical Site 33, Jerusalem, Israel
- Japan (6):
  - Clinical Site 34, Chiba
  - Clinical Site 35, Ishikawa
  - Clinical Site 36, Osaka
  - Clinical Site 37, Tochigi
  - Clinical Site 38, Tokyo
  - Clinical Site 39, Tokyo
- Mexico (3):
  - Clinical Site 41, Tlalpan, Mexico DF
  - Clinical Site 42, Cuernavaca, Morelos
  - Clinical Site 40, Mexico City
- New Zealand (3):
  - Clinical Site 44, Auckland
  - Clinical Site 43, Auckland
  - Clinical Site 45, Christchurch
- Clinical Site 46, Muscat, Oman
- Clinical Site 47, Lodz, Poland
- Serbia (2):
  - Clinical Site 48, Belgrade
  - Clinical Site 49, Niš
- Clinical Site 50, Singapore, Singapore
- South Korea (2):
  - Clinical Site 51, Gwangju
  - Clinical Site 52, Seoul
- Spain (4):
  - Clinical Site 53, A Coruña
  - Clinical Site 54, Granada
  - Clinical Site 55, Madrid
  - Clinical Site 56, Santiago de Compostela
- Turkey (Türkiye) (2):
  - Clinical Site 58, Melikgazi, Kayseri
  - Clinical Site 57, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watts GF, Rosenson RS, Hegele RA, Goldberg IJ, Gallo A, Mertens A, Baass A, Zhou R, Muhsin M, Hellawell J, Leeper NJ, Gaudet D; PALISADE Study Group. Plozasiran for Managing Persistent Chylomicronemia and Pancreatitis Risk. N Engl J Med. 2025 Jan 9;392(2):127-137. doi: 10.1056/NEJMoa2409368. Epub 2024 Sep 2. PMID 39225259
- See also: Expanded access record — https://clinicaltrials.gov/study/NCT06796426

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the 12-month Randomized Period, participants who successfully passed eligibility requirements at screening enrolled in parallel cohorts, with participants randomly assigned 2:1:2:1 to plozasiran 25 mg, volume-matched placebo, plozasiran 50 mg and volume-matched placebo, respectively.
  Results data is presented for the Randomized Period; per protocol, placebo arms were pooled for this analysis. An Open-label Extension Period is ongoing.
Groups:
- Placebo (Pooled): Randomized Period: volume-matched placebo every 3 months (Q3M) for a total of 4 doses.
  Open-label Period: plozasiran 25 mg or 50 mg (Part A), then 25 mg (Part B) Q3M for a total of 8 doses.
- ARO-APOC3 (Plozasiran) 50 mg: Randomized Period: plozasiran 50 mg Q3M for a total of 4 doses.
  Open-label Period: plozasiran 50 mg (Part A), then 25 mg (Part B) Q3M for a total of 8 doses.
Period: Overall Study
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Started (Randomized) | 25 | 26 | 24
Completed (Completed 12-month treatment in Randomized Period) | 19 | 23 | 22
Not Completed | 6 | 3 | 2
Not completed — Due to acute pancreatitis | 3 | 0 | 0
Not completed — Due to other adverse event | 0 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Other, not specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Pooled): Randomized Period: volume-matched placebo Q3M for a total of 4 doses.
  Open-label Period: plozasiran 25 mg or 50 mg (Part A), then 25 mg (Part B) Q3M for a total of 8 doses.
- Total: Total of all reporting groups
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg | Total
Number analyzed (Participants) | 25 | 26 | 24 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (13.93) | 47.9 (14.41) | 42.6 (10.85) | 46.0 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 13 | 38
  Male | 14 | 12 | 11 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 24 | 26 | 22 | 72
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 19 | 17 | 55
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 4 | 7 | 5 | 16
  Other, not specified | 2 | 0 | 1 | 3
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 2271.91 (1141.426) | 2349.53 (1374.542) | 2491.45 (1523.200) | 2369.07 (1337.965)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline at Month 10 in Fasting Triglycerides (TG)
Time Frame: Baseline, Month 10
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. Participants with an assessment at baseline and Month 10.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage change | -17.1 [-49.1 to 47.0] | -80.1 [-89.9 to -61.0] | -77.6 [-87.7 to -48.6]
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = -58.7, 95% CI 2-sided [-89.6 to -27.9] — Hodges-Lehmann method was used to estimate the median difference (location shift) and its corresponding 95% confidence interval for percent changes between plozasiran doses and placebo (pooled)
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0002, Wilcoxon rank-sum test; Median Difference (Final Values) = -52.5, 95% CI 2-sided [-83.1 to -21.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0002, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment

2. Secondary Outcome: Percent Change From Baseline in Fasting TG at Month 10 and Month 12 (Averaged)
Time Frame: Baseline, Month 10, Month 12
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. Participants with an assessment at baseline and Months 10 and 12.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage change | -2.6 [-45.0 to 33.3] | -77.7 [-89.0 to -59.2] | -71.0 [-86.7 to -52.6]
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = -59.6, 95% CI 2-sided [-91.6 to -27.5] — Hodges-Lehmann method was used to estimate the median difference (location shift) and its corresponding 95% CI for percent changes between plozasiran doses and placebo (pooled)
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0007, Wilcoxon rank-sum test; Median Difference (Final Values) = -50.8, 95% CI 2-sided [-83.5 to -18.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0007, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment

3. Secondary Outcome: Percent Change From Baseline in Apolipoprotein C-III (APOC3) at Month 10
Time Frame: Baseline, Month 10
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage change | -1.25 [-16.59 to 26.46] | -92.95 [-97.58 to -87.86] | -96.20 [-97.71 to -89.88]
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = -90.48, 95% CI 2-sided [-108.29 to -72.67] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = -93.40, 95% CI 2-sided [-109.38 to -77.42] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p < 0.0001, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment

4. Secondary Outcome: Percent Change From Baseline in Fasting APOC3 at Month 12
Time Frame: Baseline, Month 12
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. Participants with an assessment at baseline and Month 12.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage change | 7.69 [-33.65 to 31.28] | -89.30 [-93.84 to -80.24] | -87.73 [-93.01 to -78.70]
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = -86.95, 95% CI 2-sided [-112.93 to -60.96] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p < 0.0001, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = -87.48, 95% CI 2-sided [-112.42 to -62.54] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p < 0.0001, Holm method — The adjusted p-value was calculated using the Holm method for multiplicity adjustment

5. Secondary Outcome: Percentage of Participants With Positively Adjudicated Events of Acute Pancreatitis (Randomized Period)
Description: All adverse events (AEs) and serious adverse events (SAEs) reported by the Investigator during the study that are consistent with an event of acute pancreatitis will be adjudicated by a blinded, independent committee according to the 2013 Atlanta definition meeting 2 of the following 3 criteria:
  1. Abdominal pain consistent with acute pancreatitis (acute onset of a persistent, severe, epigastric pain often radiating to the back)
  2. Serum lipase activity (or amylase activity) ≥3 times the upper limit of normal (×ULN)
  3. Characteristic findings of acute pancreatitis on contrast-enhanced computed tomography (CECT), magnetic resonance imaging (MRI), or transabdominal ultrasonography.
Time Frame: From first dose of study drug through Month 12 (Randomized Period)
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. The Statistical Analysis Plan pre-specified that the ARO-APOC3 25 mg and 50 mg groups were to be pooled together to be compared with placebo for the Randomized Period.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (Pooled): Randomized Period: volume-matched placebo Q3M for a total of 4 doses.
- ARO-APOC3 (Plozasiran) Pooled: Randomized Period: plozasiran 25 mg or 50 mg Q3M for a total of 4 doses.
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) Pooled
Number analyzed (Participants) | 25 | 50
percentage of participants | 20.0 | 4.0
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) Pooled; Test type: Superiority; p = 0.0292, Cochran-Mantel-Haenszel — Odds ratio, 95% confidence interval (CI), and P-value were based on Cochran-Mantel-Haenszel (CMH) test stratified by baseline triglyceride category; Odds Ratio (OR) = 0.169, 95% CI 2-sided [0.030 to 0.942]

6. Secondary Outcome: Percentage of Participants With Positively Adjudicated Events of Acute Pancreatitis (Open-Label Period)
Description: as for outcome 5
Time Frame: From first dose of study drug through Month 36 (Open-Label Period)
Reporting Status: Not Posted, anticipated posting 2027-04

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Month 10
Time Frame: Baseline, Month 10
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. A pattern-mixture model is used as the imputation method for the missing values of Month 10 in fasting non-HDL-Cs.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 25 | 26 | 24
percentage change | 3.67 (9.454) | -38.69 (7.980) | -36.12 (8.351)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p = 0.0007, ANCOVA — ANCOVA with Pattern-mixture Model; Least squares (LS) mean difference = -42.36, 95% CI 2-sided [-66.70 to -18.01], Standard Error of Mean 12.412
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0018, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = -39.79, 95% CI 2-sided [-64.72 to -14.87], Standard Error of Mean 12.706

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Month 12
Time Frame: Baseline, Month 12
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. A pattern-mixture model is used as the imputation method for the missing values of Month 12 in fasting non-HDL-Cs.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 25 | 26 | 24
percentage change | 6.72 (9.373) | -38.16 (7.928) | -25.48 (8.368)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p = 0.0003, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = -44.88, 95% CI 2-sided [-68.86 to -20.89], Standard Error of Mean 12.230
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0114, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = -32.19, 95% CI 2-sided [-57.13 to -7.25], Standard Error of Mean 12.713

9. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Month 10
Time Frame: Baseline, Month 10
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. A pattern-mixture model is used as the imputation method for the missing values of Month 10 in fasting HDL-Cs.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 25 | 26 | 24
percentage change | 2.89 (12.281) | 65.48 (11.485) | 72.02 (12.263)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p = 0.0002, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = 62.60, 95% CI 2-sided [29.68 to 95.52], Standard Error of Mean 16.796
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = 69.14, 95% CI 2-sided [34.85 to 103.42], Standard Error of Mean 17.492

10. Secondary Outcome: Percent Change From Baseline in HDL-C at Month 12
Time Frame: Baseline, Month 12
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. A pattern-mixture model is used as the imputation method for the missing values of Month 12 in fasting HDL-Cs.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 25 | 26 | 24
percentage change | 20.61 (17.249) | 61.90 (14.462) | 74.52 (15.775)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p = 0.0669, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = 41.28, 95% CI 2-sided [-2.88 to 85.44], Standard Error of Mean 22.520
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0256, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = 53.90, 95% CI 2-sided [6.60 to 101.21], Standard Error of Mean 24.119

11. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 25 | 26 | 24
percentage change | 0.72 (15.962) | -61.50 (14.334) | -45.38 (14.542)
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Test type: Superiority; p = 0.0036, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = -62.22, 95% CI 2-sided [-104.11 to -20.32], Standard Error of Mean 21.356
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Test type: Superiority; p = 0.0338, ANCOVA — ANCOVA with Pattern-mixture Model; LS mean difference = -46.10, 95% CI 2-sided [-88.65 to -3.54], Standard Error of Mean 21.693

12. Secondary Outcome: Percentage of Participants Achieving Fasting TG of <500, 880, and 1000 mg/dL at Month 10
Time Frame: Month 10
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. Observed cases.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage of participants
  <500 mg/dL (<5.6 mmol/L) | 5.3 | 50.0 | 45.5
  <880 mg/dL (<9.9 mmol/L) | 21.1 | 75.0 | 54.5
  <1000 mg/dL (<11.3 mmol/L) | 31.6 | 83.3 | 68.2
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Number of participants with triglycerides <500 mg/dL (<5.6 mmol/L); Test type: Superiority; p = 0.0066, Regression, Logistic — The odds ratio, corresponding 95% CI and p-value are based on a logistic regression model with treatment group, and baseline triglyceride level as a covariate; Odds Ratio (OR) = 21.120, 95% CI 2-sided [2.343 to 190.405]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Number of participants with triglycerides <500 mg/dL (<5.6 mmol/L); Test type: Superiority; p = 0.0106, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 17.953, 95% CI 2-sided [1.960 to 164.414]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Number of participants with triglycerides <880 mg/dL (<9.9 mmol/L); Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 15.448, 95% CI 2-sided [3.280 to 72.762]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Number of participants with triglycerides <880 mg/dL (<9.9 mmol/L); Test type: Superiority; p = 0.0194, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 5.708, 95% CI 2-sided [1.325 to 24.596]
Statistical Analysis 5: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Number of participants with triglycerides <1000 mg/dL (<11.3 mmol/L); Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 20.838, 95% CI 2-sided [3.737 to 116.182]
Statistical Analysis 6: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Number of participants with triglycerides <1000 mg/dL (<11.3 mmol/L); Test type: Superiority; p = 0.0086, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 7.640, 95% CI 2-sided [1.676 to 34.830]

13. Secondary Outcome: Percentage of Participants Achieving Fasting TG of <500, 880, and 1000 mg/dL at Month 12
Time Frame: Month 12
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage of participants
  <500 mg/dL (<5.6 mmol/L) | 10.5 | 45.8 | 40.9
  <880 mg/dL (<9.9 mmol/L) | 26.3 | 75.0 | 59.1
  <1000 mg/dL (<11.3 mmol/L) | 26.3 | 75.0 | 63.6
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Number of participants with triglycerides <500 mg/dL (<5.6 mmol/L); Test type: Superiority; p = 0.0131, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 9.097, 95% CI 2-sided [1.589 to 52.074]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Number of participants with triglycerides <500 mg/dL (<5.6 mmol/L); Test type: Superiority; p = 0.0257, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 7.435, 95% CI 2-sided [1.275 to 43.360]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Number of participants with triglycerides <880 mg/dL (<9.9 mmol/L); Test type: Superiority; p = 0.0014, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 11.195, 95% CI 2-sided [2.553 to 49.096]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Number of participants with triglycerides <880 mg/dL (<9.9 mmol/L); Test type: Superiority; p = 0.0223, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 5.166, 95% CI 2-sided [1.263 to 21.131]
Statistical Analysis 5: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Number of participants with triglycerides <1000 mg/dL (<11.3 mmol/L); Test type: Superiority; p = 0.0013, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 11.623, 95% CI 2-sided [2.612 to 51.726]
Statistical Analysis 6: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Number of participants with triglycerides <1000 mg/dL (<11.3 mmol/L); Test type: Superiority; p = 0.0102, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 6.640, 95% CI 2-sided [1.568 to 28.119]

14. Secondary Outcome: Percentage of Participants Achieving ≥40% and ≥70% Reduction From Baseline in Fasting TG at Month 10
Time Frame: Baseline, Month 10
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 19 | 24 | 22
percentage of participants
  ≥40% reduction from baseline fasting triglycerides | 26.3 | 95.8 | 86.4
  ≥70% reduction from baseline fasting triglycerides | 10.5 | 66.7 | 54.5
Statistical Analysis 1: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Percentage of participants achieving ≥40% reduction from baseline fasting triglycerides; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 65.020, 95% CI 2-sided [6.791 to 622.535]
Statistical Analysis 2: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Percentage of participants achieving ≥40% reduction from baseline fasting triglycerides; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 17.440, 95% CI 2-sided [3.518 to 86.446]
Statistical Analysis 3: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 25 mg; Percentage of participants achieving ≥70% reduction from baseline fasting triglycerides; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 18.262, 95% CI 2-sided [3.302 to 100.991]
Statistical Analysis 4: Comparison: Placebo (Pooled) vs ARO-APOC3 (Plozasiran) 50 mg; Percentage of participants achieving ≥70% reduction from baseline fasting triglycerides; Test type: Superiority; p = 0.0057, Regression, Logistic — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 11.109, 95% CI 2-sided [2.015 to 61.235]

15. Secondary Outcome: Change From Baseline in Fasting TG Over Time
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: Full Analysis Set: all randomized participants regardless of adherence to the treatment, analyzed according to the treatment assigned at randomization. Participants with an assessment at baseline and given timepoint.
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- ARO-APOC3 (Plozasiran) 25 mg: Randomized Period: plozasiran 25 mg Q3M for a total of 4 doses.
- ARO-APOC3 (Plozasiran) 50 mg: Randomized Period: plozasiran 50 mg Q3M for a total of 4 doses.
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 24 | 25 | 23
mg/dL
  Change at Month 1: number analyzed (Participants) | 24 | 25 | 22
  Change at Month 1 | 180.81 (247.835) | -1898.79 (205.603) | -1759.36 (277.758)
  Change at Month 2: number analyzed (Participants) | 23 | 25 | 22
  Change at Month 2 | -203.67 (195.740) | -1519.38 (203.397) | -1481.57 (218.704)
  Change at Month 3: number analyzed (Participants) | 23 | 25 | 22
  Change at Month 3 | 392.98 (320.073) | -1177.43 (212.134) | -1478.94 (276.681)
  Change at Month 4: number analyzed (Participants) | 23 | 24 | 23
  Change at Month 4 | -248.76 (198.553) | -1521.25 (291.471) | -1810.31 (245.695)
  Change at Month 5: number analyzed (Participants) | 23 | 24 | 23
  Change at Month 5 | -213.43 (216.851) | -1613.90 (176.086) | -1689.31 (330.096)
  Change at Month 6: number analyzed (Participants) | 22 | 24 | 22
  Change at Month 6 | -276.07 (205.490) | -1566.97 (201.610) | -1325.13 (215.809)
  Change at Month 7: number analyzed (Participants) | 23 | 24 | 22
  Change at Month 7 | 324.98 (319.233) | -1842.65 (210.671) | -1691.87 (285.252)
  Change at Month 8: number analyzed (Participants) | 22 | 25 | 23
  Change at Month 8 | 188.62 (271.286) | -1537.57 (190.088) | -1133.96 (279.984)
  Change at Month 9: number analyzed (Participants) | 19 | 25 | 22
  Change at Month 9 | -119.48 (226.547) | -1413.87 (232.426) | -1650.75 (329.600)
  Change at Month 10: number analyzed (Participants) | 19 | 24 | 22
  Change at Month 10 | -248.35 (233.539) | -1819.82 (227.632) | -1740.20 (293.567)
  Change at Month 11: number analyzed (Participants) | 18 | 22 | 21
  Change at Month 11 | 173.14 (336.713) | -1810.57 (296.726) | -1507.08 (203.964)
  Change at Month 12: number analyzed (Participants) | 19 | 24 | 22
  Change at Month 12 | -50.32 (273.674) | -1637.18 (274.479) | -1485.30 (339.662)

16. Secondary Outcome: Percent Change From Baseline in Fasting TG Over Time
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 15
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 24 | 25 | 23
percentage change
  Percent Change at Month 1: number analyzed (Participants) | 24 | 25 | 22
  Percent Change at Month 1 | 13.21 (14.003) | -81.43 (2.854) | -68.21 (5.390)
  Percent Change at Month 2: number analyzed (Participants) | 23 | 25 | 22
  Percent Change at Month 2 | -7.30 (10.375) | -69.33 (5.119) | -62.96 (5.940)
  Percent Change at Month 3: number analyzed (Participants) | 23 | 25 | 22
  Percent Change at Month 3 | 14.66 (12.028) | -57.13 (7.424) | -60.94 (6.761)
  Percent Change at Month 4: number analyzed (Participants) | 23 | 24 | 23
  Percent Change at Month 4 | -1.74 (8.861) | -68.27 (8.795) | -71.91 (5.076)
  Percent Change at Month 5: number analyzed (Participants) | 23 | 24 | 23
  Percent Change at Month 5 | -9.23 (9.561) | -71.96 (5.052) | -60.41 (10.796)
  Percent Change at Month 6: number analyzed (Participants) | 22 | 24 | 22
  Percent Change at Month 6 | -6.18 (12.679) | -68.08 (4.884) | -56.30 (6.317)
  Percent Change at Month 7: number analyzed (Participants) | 23 | 24 | 22
  Percent Change at Month 7 | 21.45 (15.235) | -77.44 (4.082) | -65.88 (5.863)
  Percent Change at Month 8: number analyzed (Participants) | 22 | 25 | 23
  Percent Change at Month 8 | 14.98 (13.745) | -68.35 (4.805) | -47.77 (11.563)
  Percent Change at Month 9: number analyzed (Participants) | 19 | 25 | 22
  Percent Change at Month 9 | 4.08 (12.059) | -55.32 (8.363) | -62.72 (7.369)
  Percent Change at Month 10: number analyzed (Participants) | 19 | 24 | 22
  Percent Change at Month 10 | -8.74 (11.466) | -74.45 (4.135) | -66.53 (5.951)
  Percent Change at Month 11: number analyzed (Participants) | 18 | 22 | 21
  Percent Change at Month 11 | 10.40 (16.139) | -68.39 (6.776) | -63.83 (6.143)
  Percent Change at Month 12: number analyzed (Participants) | 19 | 24 | 22
  Percent Change at Month 12 | 0.93 (14.858) | -67.69 (5.985) | -50.60 (14.269)

17. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and/or Serious Adverse Events (SAEs; Randomized Period)
Description: AE: any untoward medical occurrence which does not necessarily have to have a causal relationship with treatment. Treatment-emergent AEs (TEAEs): AEs with onset after administration of the study drug, or when a preexisting medical condition increases in severity or frequency after study drug administration. SAE: AE that fulfills one or more of the following: results in death; is immediately life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above. Severity was reported as: mild, moderate, severe, life threatening, death.
Time Frame: From first dose of study drug through Month 12 (Randomized Period)
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug, analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
Number analyzed (Participants) | 25 | 26 | 24
Participants
  All TEAEs | 20 | 23 | 20
  Treatment-related TEAEs | 6 | 7 | 8
  Serious TEAEs | 7 | 5 | 2
  TEAEs leading to study drug discontinuation | 0 | 2 | 1
  TEAEs leading to study termination | 0 | 2 | 1
  TEAEs of clinical interest | 1 | 4 | 2
  Any TEAE by maximum severity: Mild | 5 | 13 | 13
  Any TEAE by maximum severity: Moderate | 10 | 7 | 4
  Any TEAE by maximum severity: Severe | 5 | 2 | 3
  Any TEAE by maximum severity: Life Threatening | 0 | 1 | 0
  Any TEAE by maximum severity: Death | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Treatment-Emergent AEs and/or SAEs (Open-Label Period)
Description: as for outcome 17
Time Frame: From first dose of open-label study drug through Month 36 (Open-Label Period)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Screening through Month 12 (Randomized Period)
Arm/Group | Placebo (Pooled) | ARO-APOC3 (Plozasiran) 25 mg | ARO-APOC3 (Plozasiran) 50 mg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 7/25 | 5/26 | 2/24
Other Adverse Events (participants affected / at risk) | 17/25 | 21/26 | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pooled) (N=25) | ARO-APOC3 (Plozasiran) 25 mg (N=26) | ARO-APOC3 (Plozasiran) 50 mg (N=24)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 3 | 2 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 3 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pooled) (N=25) | ARO-APOC3 (Plozasiran) 25 mg (N=26) | ARO-APOC3 (Plozasiran) 50 mg (N=24)
Palpitations (Cardiac disorders) | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 7
Nausea (Gastrointestinal disorders) | 2 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2
Fatigue (General disorders) | 2 | 1 | 2
Injection site pain (General disorders) | 1 | 2 | 1
Injection site reaction (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 1 | 5 | 7
Nasopharyngitis (Infections and infestations) | 4 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 3 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 3 | 5
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05089084/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT05089084/SAP_002.pdf